CLINICAL TRIAL: NCT01030536
Title: A Phase 1/2 Study of CAT-8015 in Adult Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma and Chronic Lymphocytic Leukemia
Brief Title: Safety Study of CAT-8015 to Treat Advanced B-cell Non-Hodgkin Lymphoma and Chronic Lymphocytic Leukemia (NHL or CLL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP218; NCT01086644 (obsolete NCT alias)
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-03

CONDITIONS: Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
Keywords: NHL; CLL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — immunotoxin HA22

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- CAT-8015 20 microgram per kilogram (mcg/kg) (Experimental): Participants will receive 20 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle. Dose escalation is to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level are possible if an MTD or OBD is not reached by 60 mcg/kg.
  Interventions: Drug: CAT-8015 20 mcg/kg
- CAT-8015 30 mcg/kg (Experimental): Participants will receive 30 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle. Dose escalation is to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level are possible if an MTD or OBD is not reached by 60 mcg/kg.
  Interventions: Drug: CAT-8015 30 mcg/kg
- CAT-8015 40 mcg/kg (Experimental): Participants will receive 40 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle. Dose escalation is to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level are possible if an MTD or OBD is not reached by 60 mcg/kg.
  Interventions: Drug: CAT-8015 40 mcg/kg
- CAT-8015 50 mcg/kg (Experimental): Participants will receive 50 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle. Dose escalation is to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level are possible if an MTD or OBD is not reached by 60 mcg/kg.
  Interventions: Drug: CAT-8015 50 mcg/kg
- CAT-8015 60 mcg/kg (Experimental): Participants will receive 60 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle. Dose escalation is to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level are possible if an MTD or OBD is not reached by 60 mcg/kg.
  Interventions: Drug: CAT-8015 60 mcg/kg

INTERVENTIONS:
Drug: CAT-8015 20 mcg/kg — Participants will receive 20 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle.
  Arms: CAT-8015 20 microgram per kilogram (mcg/kg)
Drug: CAT-8015 30 mcg/kg — Participants will receive 30 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle.
  Arms: CAT-8015 30 mcg/kg
Drug: CAT-8015 40 mcg/kg — Participants will receive 40 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle.
  Arms: CAT-8015 40 mcg/kg
Drug: CAT-8015 50 mcg/kg — Participants will receive 50 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle.
  Arms: CAT-8015 50 mcg/kg
Drug: CAT-8015 60 mcg/kg — Participants will receive 60 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle.
  Arms: CAT-8015 60 mcg/kg

SUMMARY:
The primary objectives of this study are to determine the maximum tolerated dose (MTD) or optimal biologic dose (OBD) and safety profile of CAT-8015 in participants with relapsed or refractory advanced B-cell NHL (diffuse large B-cell lymphoma [DLBCL], follicular lymphoma [FL], mantle cell lymphoma [MCL]) or CLL.

DETAILED DESCRIPTION:
To determine the maximum tolerated dose (MTD) or optimal biologic dose (OBD) of CAT-8015 in participants with relapsed or refractory advanced B-cell NHL (DLBCL, FL, MCL) or CLL.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization
* Participants must have histologically confirmed B-cell CLL, including small lymphocytic lymphoma (SLL), DLBCL, MCL, or FL
* B-cell NHL: a) Have previous confirmation of B-cell NHL b) Participants with DLBCL or MCL, must have relapsed or refractory disease after at least one prior regimen containing rituximab, either alone or in combination, and be ineligible for any available standard line of therapy known to be life-prolonging or life-saving c) Participants with FL, must have relapsed or refractory disease after at least two prior regimens, one of which included rituximab, either alone or in combination, and be ineligible for any available standard line of therapy known to be life-prolonging or life-saving d) Have measurable disease (at least one lesion greater than or equal to (≥) 20 millimeter (mm) in one dimension or ≥ 15 mm in two dimensions as measured by conventional or high resolution [spiral] computed tomography e) Not be a candidate for a hematopoietic stem cell (HSC) or bone marrow transplant
* B-cell CLL: a) Have previous confirmation of B-cell CLL with a characteristic immunophenotype by flow cytometry b) Have relapsed or refractory disease after at least 2 prior lines of treatment, at least 1 of which must have contained rituximab and be ineligible for any available standard line of therapy known to be life-prolonging or life-saving c) Not be a candidate for an HSC or BM transplant d) Have symptomatic disease that requires treatment
* Karnofsky Performance Status ≥ 70
* Life expectancy of ≥ 12 weeks
* Toxicities from previous cancer therapies must have recovered to Grade less than (<) 2
* Adequate hematological function defined as: a) Hemoglobin ≥ 9 g/dL b) Absolute neutrophil count ≥ 1500/mm^3 c) Platelet count ≥ 75,000/mm^3
* Prothrombin time-International Normalized Ratio/Partial thromboplastin time less than or equal to (≤) 1.5 × upper limit of normal (ULN), or for participants on anticoagulation therapy, status within therapeutic range
* Women of non-child-bearing potential or using effective contraception
* Male participants with partners of child-bearing potential must be surgically sterile or use a contraceptive method

Exclusion Criteria:

* Any available standard line of therapy known to be life-prolonging or life-saving
* Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic, or hormonal therapy for treatment of cancer
* For CLL participants only, rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy
* History of allergy or reaction to any component of the CAT-8015
* Receipt of any chemotherapy or small molecule targeted therapy or any biological- or immunological-based therapies for leukemia or lymphoma within 6 weeks
* Prior radiation therapy will not be excluded, providing the volume of bone marrow treated is less than 25 percent
* Any history of prior pseudomonas-exotoxin immunotoxin administration including CAT-8015, CAT-3888, or LMB-2
* History of other invasive malignancy within 5 years, with some exceptions
* Evidence of significant active infection requiring antimicrobial, antifungal, antiparasitic or antiviral therapy or for which other supportive care is given
* Autologous stem cell transplantation within 6 months prior to study entry
* Allogenic stem cell transplantation or any other organ transplant
* HIV-positive or AIDS, Hepatitis B or hepatitis C infection as defined by seropositive for hepatitis B (HBsAg) or hepatitis C and elevated liver transaminases
* Use of immunosuppressive medication other than steroids within 7 days, use of systemic steroids within 7 days before the first dose of CAT-8015 (inhaled and topical corticosteroids are permitted). Participants may take replacement doses of steroids (defined as ≤ 30 mg/day hydrocortisone or the equivalent) if on a stable dose for at least 2 weeks prior to the first dose of CAT-8015
* Documented current central nervous system involvement by leukemia or lymphoma
* Pregnancy or lactation, other severe, concurrent diseases
* Concurrent enrollment in another clinical study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-02-15 (Actual); Primary Completion 2013-03-04 (Actual); Study Completion 2013-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramy Ibrahim, M.D., Study Director — MedImmune LLC
Locations (8):
- United States (7):
  - Research Site, Los Angeles, California
  - Research Site, Indianapolis, Indiana
  - Research Site, Bethesda, Maryland
  - Research Site, Las Vegas, Nevada
  - Research Site, Charleston, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Temple, Texas
- Research Site, Lodz, Poland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was started on 15 Feb 2010 and was terminated on 12 Sep 2012. The Product Development Team authorized early termination of this study due to prioritization of resources and the need to prioritize allocation of investigational product across the studies in the moxetumomab pasudotox clinical development program.
Pre-assignment Details: A total of 30 participants were screened and enrolled, of them 7 were failed screening. Twenty three participants were enrolled and assigned to treatment at 6 sites in the United States.
Groups:
- CAT-8015 20 Microgram Per Kilogram (mcg/kg): Participants received 20 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle. Dose escalation was to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level were possible if an MTD or OBD was not reached by 60 mcg/kg.
- CAT-8015 30 Microgram Per Kilogram (mcg/kg): Participants received 30 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle. Dose escalation was to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level were possible if an MTD or OBD was not reached by 60 mcg/kg.
- CAT-8015 40 Microgram Per Kilogram (mcg/kg): Participants received 40 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle. Dose escalation was to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level were possible if an MTD or OBD was not reached by 60 mcg/kg.
- CAT-8015 50 Microgram Per Kilogram (mcg/kg): Participants received 50 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle. Dose escalation was to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level were possible if an MTD or OBD was not reached by 60 mcg/kg.
- CAT-8015 60 Microgram Per Kilogram (mcg/kg): Participants received 60 mcg/kg Moxetumomab pasudotox (CAT-8015) as an intravenous (IV) infusion over 30 minutes on Days 1, 3, and 5 of every 28-day cycle. Dose escalation was to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level were possible if an MTD or OBD was not reached by 60 mcg/kg.
Period: Overall Study
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Started | 7 | 6 | 6 | 3 | 1
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 6 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — undefined | 1 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 3 | 1 | 0 | 1
Not completed — Progressive disease | 6 | 2 | 3 | 2 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg) | Total
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 1 | 23
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 63.4 (8.7) | 53.7 (16.9) | 63.5 (10.0) | 52.3 (14.6) | 66.0 (NA) — Data was not calculated | 59.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 0 | 1 | 4
  Male | 5 | 5 | 6 | 3 | 0 | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD reflects highest dose of drug that did not cause an unacceptable side effect (= Dose Limiting Toxicity [DLT]) in more than 30 percent (%) of participants.
Time Frame: Day 1 to end of Cycle 1 (approximately 28 days)
Population: Evaluable Population for DLT included all participants enrolled in the dose-escalation phase who received at least one full cycle of moxetumomab pasudotox and completed safety follow-up through the DLT evaluation period or experienced any DLT.
Measure: Number; unit: mcg/Kg
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 1
mcg/Kg | NA — Data was not reported as MTD was not reached in the specified arm group. | NA — Data was not reported as MTD was not reached in the specified arm group. | NA — Data was not reported as MTD was not reached in the specified arm group. | NA — Data was not reported as MTD was not reached in the specified arm group. | NA — Data was not reported as MTD was not reached in the specified arm group.

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Any Grade 3 or greater, non-hematological toxicity (including capillary leak syndrome [CLS] and thrombotic microangiopathy/ hemolytic uremic syndrome (HUS), Grade 3 or higher treatment-related hematologic toxicities and only ≥ Grade 3 thrombotic microangiopathy /HUS constituted a DLT with few exceptions.
Time Frame: Day 1 to end of Cycle 1 (approximately 28 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 1
Participants | 0 | 2 | 1 | 0 | 1

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: Treatment-emergent adverse event (TEAEs) were defined as events that occur following the first injection of study treatment, or that started prior to the first injection and worsened during treatment. An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An Serious Adverse Event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent adverse events were defined as adverse events/serious adverse events that started or worsened after the study drug treatment.
Time Frame: From Screening (Day -28) to Post Therapy Day 30
Population: Safety Population included all participants who received moxetumomab pasudotox. The safety population was used to evaluate baseline characteristics as well as all endpoints for safety.
Measure: Count of Participants; unit: Participants
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 1
Participants
  TEAEs | 7 | 6 | 6 | 3 | 1
  TESAEs | 0 | 3 | 2 | 0 | 1

4. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Recorded as Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse event (TEAEs) were defined as events that occur following the first injection of study treatment, or that started prior to the first injection and worsened during treatment. An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent adverse events were defined as adverse events/serious adverse events that started or worsened after the study drug treatment.
Time Frame: From Screening (Day -28) to Post Therapy Day 30
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 1
Participants
  Anaemia | 0 | 3 | 3 | 0 | 1
  Neutrophil count decreased | 1 | 0 | 0 | 1 | 1
  Neutropenia | 1 | 1 | 0 | 0 | 0
  Platelet count decreased | 0 | 0 | 1 | 0 | 1
  Thrombocytopenia | 0 | 2 | 0 | 0 | 0
  Leukocytosis | 0 | 1 | 0 | 0 | 0
  Hypoalbuminaemia | 2 | 1 | 2 | 0 | 1
  Hypertriglyceridaemia | 0 | 3 | 0 | 1 | 1
  Hyponatraemia | 0 | 1 | 3 | 0 | 1
  Alanine aminotransferase increased | 1 | 1 | 0 | 1 | 1
  Blood creatinine increased | 1 | 2 | 0 | 0 | 1
  Hypernatraemia | 2 | 0 | 1 | 0 | 1
  Hypocalcaemia | 0 | 1 | 2 | 0 | 1
  Aspartate aminotransferase increased | 1 | 1 | 0 | 1 | 0
  Hypokalaemia | 0 | 0 | 1 | 1 | 1
  Blood alkaline phosphatase increased | 0 | 0 | 0 | 1 | 1
  Hypercalcaemia | 0 | 1 | 0 | 0 | 1
  Hyperglycaemia | 0 | 1 | 1 | 0 | 0
  Hyperkalaemia | 0 | 1 | 1 | 0 | 0
  Hyperuricaemia | 1 | 0 | 0 | 0 | 1
  Hypophosphataemia | 0 | 0 | 1 | 1 | 0
  Blood albumin decreased | 1 | 0 | 0 | 0 | 0
  Blood bicarbonate increased | 0 | 0 | 0 | 0 | 1
  Blood bilirubin increased | 1 | 0 | 0 | 0 | 0
  Blood triglycerides increased | 0 | 1 | 0 | 0 | 0
  Haptoglobin decreased | 0 | 0 | 0 | 0 | 1
  Hyperchlorhydria | 0 | 0 | 1 | 0 | 0
  Hyperlipidaemia | 0 | 0 | 1 | 0 | 0
  Hypermagnesaemia | 0 | 0 | 0 | 0 | 1
  Hematuria | 0 | 1 | 1 | 0 | 1

5. Primary Outcome: Number of Participants With Vital Signs Abnormalities Recorded as Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 4
Time Frame: From Screening (Day -28) to Post Therapy Day 30
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 1
Participants
  Hypotension | 1 | 1 | 1 | 0 | 1
  Hypertension | 0 | 2 | 1 | 0 | 0
  Pyrexia | 0 | 1 | 1 | 0 | 0
  Weight Increased | 1 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities Recorded as Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 4
Time Frame: From Screening (Day -28) to Post Therapy Day 30
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 1
Participants
  Sinus Tachycardia | 0 | 1 | 0 | 0 | 0
  ECG QT Prolonged | 2 | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants With Complete Response (CR)
Description: The CR rate was defined as the percentage of participants who had achieved CR based on both the evaluable population for efficacy.
Time Frame: Baseline (Day 1) until Final Study Visit Post Therapy (up to 2 year after the last participant begins study drug treatment)
Population: Evaluable Population for efficacy included all participants who received any moxetumomab pasudotox treatment and completed at least one post-baseline disease assessment. The Evaluable Population for efficacy was used to evaluate the endpoints for the efficacy profile.
Measure: Number; unit: Percentage of Participants
Groups:
- Chronic Lymphocytic Leukemia: Participants with Chronic Lymphocytic Leukemia were included. Moxetumomab pasudotox was administered at doses of 20, 30, 40, 50, or 60 mcg/kg on Days 1, 3, and 5 of every 28-day cycle. Dose escalation was to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level were possible if an MTD or OBD was not reached by 60mcg/kg.
- Diffuse Large B Cell Lymphoma: Participants with Diffuse Large B cell Lymphoma were included. Moxetumomab pasudotox was administered at doses of 20, 30, 40, 50, or 60 mcg/kg on Days 1, 3, and 5 of every 28-day cycle. Dose escalation was to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level were possible if an MTD or OBD was not reached by 60mcg/kg.
- Mantle Cell Lymphoma: Participants with Mantle Cell Lymphoma were included. Moxetumomab pasudotox was administered at doses of 20, 30, 40, 50, or 60 mcg/kg on Days 1, 3, and 5 of every 28-day cycle. Dose escalation was to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level were possible if an MTD or OBD was not reached by 60mcg/kg.
- Follicular Lymphoma: Participants with Follicular Lymphoma (FL) were included. Moxetumomab pasudotox was administered at doses of 20, 30, 40, 50, or 60 mcg/kg on Days 1, 3, and 5 of every 28-day cycle. Dose escalation was to be continued to the Maximum tolerated dose (MTD) or Optimal biologic dose (OBD). Subsequent dose levels with a 10 mcg/kg increase from the previous dose level were possible if an MTD or OBD was not reached by 60mcg/kg.
Arm/Group | Chronic Lymphocytic Leukemia | Diffuse Large B Cell Lymphoma | Mantle Cell Lymphoma | Follicular Lymphoma
Number analyzed (Participants) | 10 | 6 | 1 | 3
Percentage of Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Duration of Complete Response
Description: Duration of CR was measured from the first documentation of a CR to the time of relapse for the subgroup of participants with CR. Duration of CR was calculated using the Kaplan Meier method. The Evaluable Population for efficacy was used to evaluate the endpoints for the efficacy profile.
Time Frame: as for outcome 7
Population: Evaluable Population for efficacy included all participants who received any moxetumomab pasudotox treatment and completed at least one post-baseline disease assessment.
Measure: Median (Full Range); unit: Months
Arm/Group | Chronic Lymphocytic Leukemia | Diffuse Large B Cell Lymphoma | Mantle Cell Lymphoma | Follicular Lymphoma
Number analyzed (Participants) | 10 | 6 | 1 | 3
Months | NA [NA to NA] — No participants had complete response over the study period, so duration of complete response could not be assessed. | NA [NA to NA] — No participants had complete response over the study period, so duration of complete response could not be assessed. | NA [NA to NA] — No participants had complete response over the study period, so duration of complete response could not be assessed. | NA [NA to NA] — No participants had complete response over the study period, so duration of complete response could not be assessed.

9. Secondary Outcome: Percentage of Participants With Partial Response (PR)
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Chronic Lymphocytic Leukemia | Diffuse Large B Cell Lymphoma | Mantle Cell Lymphoma | Follicular Lymphoma
Number analyzed (Participants) | 10 | 6 | 1 | 3
Percentage of Participants | 10 | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: OR was defined as the percentage of participants with CR or partial response (PR).
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Chronic Lymphocytic Leukemia | Diffuse Large B Cell Lymphoma | Mantle Cell Lymphoma | Follicular Lymphoma
Number analyzed (Participants) | 10 | 6 | 1 | 3
Percentage of Participants | 10 | 0 | 0 | 0

11. Secondary Outcome: Time to Response (TTR)
Description: TTR was measured from the start of moxetumomab pasudotox administration to the first documentation of response (CR or PR) and was only assessed in participants who had achieved objective response (OR).
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Median (Full Range); unit: Months
Arm/Group | Chronic Lymphocytic Leukemia | Diffuse Large B Cell Lymphoma | Mantle Cell Lymphoma | Follicular Lymphoma
Number analyzed (Participants) | 10 | 6 | 1 | 3
Months | 0.79 [0.79 to 0.79] | NA [NA to NA] — No participants had partial or complete response, so time to response could not be assessed. | NA [NA to NA] — No participants had partial or complete response, so time to response could not be assessed. | NA [NA to NA] — No participants had partial or complete response, so time to response could not be assessed.

12. Secondary Outcome: Duration of Objective Response (DOR)
Description: DOR was measured from the first documentation of OR to the event of relapse. DOR was calculated using the Kaplan-Meier method.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Median (Full Range); unit: Months
Arm/Group | Chronic Lymphocytic Leukemia | Diffuse Large B Cell Lymphoma | Mantle Cell Lymphoma | Follicular Lymphoma
Number analyzed (Participants) | 10 | 6 | 1 | 3
Months | 7.66 [7.66 to 7.66] | NA [NA to NA] — No participants had partial or complete response, so duration of objective response could not be assessed. | NA [NA to NA] — No participants had partial or complete response, so duration of objective response could not be assessed. | NA [NA to NA] — No participants had partial or complete response, so duration of objective response could not be assessed.

13. Secondary Outcome: Duration of Stable Disease (SD)
Description: Duration of SD was defined as the time period from start of moxetumomab pasudotox administration to the event of progressive disease (PD)/relapse. Duration of SD was only calculated for the subgroup of participants with best response of CR, PR, or SD, and was calculated using the Kaplan-Meier method.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Median (Full Range); unit: Months
Arm/Group | Chronic Lymphocytic Leukemia | Diffuse Large B Cell Lymphoma | Mantle Cell Lymphoma | Follicular Lymphoma
Number analyzed (Participants) | 10 | 6 | 1 | 3
Months | 1.87 [0.79 to 8.41] | NA [NA to NA] — No participants had objective response (either complete or partial response) or stable disease, so duration of stable disease could not be assessed. | 0.95 [0.95 to 0.95] | 4.67 [3.71 to 5.62]

14. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Moxetumomab Pasudotox
Description: Maximum observed drug concentration of Moxetumomab pasudotox in plasma.
Time Frame: Pre-dose and End of infusion on Day 1, 3 and 5 of each cycle; 1, 3 and 6 hour after the end of infusion on Day 1 of each cycle
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 1
nanogram per milliliter (ng/mL) | 283 (159) | 452 (141) | 589 (366) | 769 (221) | 818 (NA) — Standard Deviation was not calculated as only one participant was evaluated

15. Secondary Outcome: Area Under Concentration-Time Curve From Dosing Extrapolated to Infinity (AUCinf) of Moxetumomab Pasudotox
Description: Area under the concentration versus time curve from zero to infinity (AUC) of Moxetumomab pasudotox in Plasma.
Time Frame: as for outcome 14
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1
hour*nanogram per milliliter (hr*ng/mL) | 1120 (928) | 1640 (682) | 2050 (1150) | 2320 (1010) | 1810 (NA) — Standard Deviation was not calculated as only one participant was evaluated

16. Secondary Outcome: Clearance (CL) of Moxetumomab Pasudotox
Description: CL of drug is rate at which drug is metabolized or eliminated by normal biological processes and is influenced by fraction of dose absorbed.
Time Frame: as for outcome 14
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliliter per hour per kilogram
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1
milliliter per hour per kilogram | 31.6 (25.5) | 22.2 (12.5) | 26.9 (18.6) | 25.2 (12.9) | 33.1 (NA) — Standard Deviation was not calculated as only one participant was evaluated

17. Secondary Outcome: Elimination Half Life (t1/2) of Moxetumomab Pasudotox
Description: Plasma decay half life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 14
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1
hour | 1.55 (1.10) | 1.87 (0.985) | 1.68 (0.726) | 1.87 (0.586) | 0.901 (NA) — Standard Deviation was not calculated as only one participant was evaluated

18. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody
Description: The moxetumomab pasudotox specific bridging assay using the Meso Scale Discovery platform was employed to detect anti-drug antibodies (ADA).
Time Frame: Baseline (Day 1) up to End of the Treatment (Last dose of Last cycle) (approximately 3 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 1
Participants | 5 | 4 | 5 | 2 | 0

19. Secondary Outcome: Number of Participants With CD22 Expression Levels
Description: CD22 Expression was analyzed using Prism® analysis. Flow cytometry was performed to quantitate the CD22 expression for the purpose of evaluating the relationship of CD22 expression with response to treatment.
Time Frame: Baseline (Day 1) up to End of the Treatment (Last dose of Last cycle) (approximately 3 years)
Population: Evaluable population for expression of CD22 on malignant cells included all participants with peripheral blood samples containing 10 or more B cells (CD19-positive cells) per cubic millimeter.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Lymphocytic Leukemia | Diffuse Large B Cell Lymphoma | Mantle Cell Lymphoma | Follicular Lymphoma
Number analyzed (Participants) | 10 | 7 | 2 | 4
Participants | 8 | 5 | 2 | 1

20. Secondary Outcome: Number of Capillary Leak Syndrome (CLS) Participants With Weight Changes, Albumin, Hypotension, Edema, Hypoxia, and Pulmonary Adverse Events (AEs)
Description: The correlation of CLS and weight changes, albumin, hypotension, edema, hypoxia, and pulmonary AEs were examined.
Time Frame: From Screening (Day -28) to Post Therapy Day 30
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 1
Participants | 1 | 0 | 1 | 0 | 0

21. Secondary Outcome: Percentage of Participants With Stable Disease (SD)
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Chronic Lymphocytic Leukemia | Diffuse Large B Cell Lymphoma | Mantle Cell Lymphoma | Follicular Lymphoma
Number analyzed (Participants) | 10 | 6 | 1 | 3
Percentage of Participants | 40.0 | 0.0 | 100.0 | 66.7

ADVERSE EVENTS:
Time Frame: From Screening (Day -28) to Post Therapy Day 30
Arm/Group | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) | CAT-8015 60 Microgram Per Kilogram (mcg/kg)
Serious Adverse Events (participants affected / at risk) | 0/7 | 3/6 | 2/6 | 0/3 | 1/1
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 6/6 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAT-8015 20 Microgram Per Kilogram (mcg/kg) (N=7) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) (N=6) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) (N=6) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) (N=3) | CAT-8015 60 Microgram Per Kilogram (mcg/kg) (N=1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAT-8015 20 Microgram Per Kilogram (mcg/kg) (N=7) | CAT-8015 30 Microgram Per Kilogram (mcg/kg) (N=6) | CAT-8015 40 Microgram Per Kilogram (mcg/kg) (N=6) | CAT-8015 50 Microgram Per Kilogram (mcg/kg) (N=3) | CAT-8015 60 Microgram Per Kilogram (mcg/kg) (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 3 (4) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 5 (6) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 4 (5) | 1 (1) | 3 (11) | 2 (3) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 2 (8) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (9) | 0 (0) | 1 (2) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (4) | 1 (1) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (5) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (7) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.